CLINICAL TRIAL: NCT00760812
Title: Effects of Parent-Implemented Intervention for Toddlers With Autism Spectrum (The ESI Study)
Brief Title: Comparing Parent-Implemented Interventions for Toddlers With Autism Spectrum Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Amy M. Wetherby, Distinguished Research Professor, Florida State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH077730 (NIH); R01MH077730 (NIH); 1R01MH077730-01A2 (NIH); 1R01MH078165-01A2 (NIH); DDTR B2-MBA (Other Grant/Funding Number: National Institute of Mental Health)
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2022-07-27 (Actual); Status verified 2014-02

CONDITIONS: Autistic Disorder
Keywords: Autism; Autism Spectrum Disorders; Pervasive Developmental Disorders; Toddlers; Intervention
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Child Development Disorders, Pervasive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ESI--Individual PII First Condition (Experimental): This group will first receive the Early Social Interaction (ESI) model individual parent-implemented intervention (PII) for 9 months, followed by the ESI model group information, education, and support (IES) intervention for 9 months.
  Interventions: Behavioral: Early Social Interaction Project- PII; Behavioral: Early Social Interaction Project- IES
- ESI--Group IES First Condition (Experimental): The group will first receive ESI group IES condition for 9 months, followed by ESI individual PII for 9 months.
  Interventions: Behavioral: Early Social Interaction Project- PII; Behavioral: Early Social Interaction Project- IES

INTERVENTIONS:
Behavioral: Early Social Interaction Project- PII — The PII is an intensive, individualized treatment that teaches parents how to support social communication skills in children with autism by embedding skills practice within everyday routines, activities, and places. Participants will have three 75-minute sessions weekly with study administrators for the first 7 months of the study. Participants will then have two sessions per week for the final 2 months of the study. Children will also practice socialization embedded in normal activities for 25 hours a week outside of study visits.
Behavioral: Early Social Interaction Project- IES — The IES intervention provides access to a support group meeting twice monthly for children with autism and their parents. The support group provides information to families and a playgroup where parents may practice intervention strategies under the supervision of study officials knowledgeable about autism spectrum disorders.

SUMMARY:
This study will compare the effectiveness of two parent-based programs for helping young children at risk of autism.

DETAILED DESCRIPTION:
Autism is a problem with normal social development and is characterized by impairments in three categories: social skills, language, and behavior. Symptoms include disinterest or inability to have normal social relationships, abnormal speech or usage of phrases, and repetitive movements or rituals; these symptoms generally emerge by 18 months of age. Autism is a spectrum disorder, meaning that its symptoms can range in severity from mild to severe. There is no cure for autism, nor is there a single known cause. There are only factors known to make it more likely for children to develop autism. These include being a male, having siblings with the disorder, having certain other disorders, or having an older father. Treatments for autism generally include therapies that help children develop social communication skills and that help structure family time and school so that parents and teachers can address particular difficulties children with autism might have. Medications may also be used to counteract anxieties or compulsive behaviors.

Research has shown that earlier interventions in children who are at risk of autism may lead to better outcomes. This study will compare two interventions for developing social communication skills in children who are at risk of autism and are between 16 and 20 months old. The parent-implemented intervention (PII) will be a more intense, individualized approach, teaching parents to embed 25 hours of social communication skills practice per week in their children's daily lives. The information, education, and support (IES) intervention will offer parents a support group and place to practice methods of helping their children learn adaptive social communication.

Participation in this study will last 18 months. Participants will be randomly assigned to first receive 9 months of either PII or IES and then receive 9 months of whichever intervention they did not receive initially. The PII intervention will involve three weekly sessions for 7 months, then two weekly sessions for 2 months. The IES intervention will involve group meetings twice monthly and offer a playground where parents can practice intervention strategies with their children. All parents will complete questionnaires about family resources and social and emotional issues before the first intervention begins, after 9 months when the intervention changes, and after 18 months when the second intervention ends. Children and parents will also be assessed once a month throughout the study on social communication, autism symptoms, developmental level, and hours spent on learned strategies or techniques outside the study visits. These assessments will involve clinical assessments of parent and child behaviors (some of which will be videotaped), tests of children's abilities, and reports by parents on strategies and techniques used outside the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of autism risk factors and a clinical diagnosis of autism spectrum disorder based on a diagnostic evaluation conducted by the project team
2. Families agree to twice monthly play group sessions for 9 months and two to three intervention sessions per week for 9 months, usually to be scheduled within workday hours
3. Families agree to monthly evaluations, videotaping of intervention sessions, and weekly or monthly video checks during the 18 months of treatment

Exclusion Criteria:

1. Child does not have normal hearing or adequate motor control to make simple actions, such as giving and reaching gestures
2. Primary language of family is not English

Ages: 16 Months to 20 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2007-04; Primary Completion 2013-05 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Child measures of autism symptoms, social communication, developmental level, and adaptive behavior | Measured before treatment, at crossover, and after treatment; some of these measures also will be taken every other month

SECONDARY OUTCOMES:
Parent report measures of family functioning, daily hassles, and treatment satisfaction | Measured before treatment, at crossover, and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Amy M. Wetherby, PhD, Principal Investigator — Florida State University; Catherine Lord, PhD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - Florida State University, Tallahassee, Florida
  - University of Michigan, Ann Arbor, Michigan

REFERENCES:
- [Derived] Wetherby AM, Guthrie W, Woods J, Schatschneider C, Holland RD, Morgan L, Lord C. Parent-implemented social intervention for toddlers with autism: an RCT. Pediatrics. 2014 Dec;134(6):1084-93. doi: 10.1542/peds.2014-0757. Epub 2014 Nov 3. PMID 25367544